CLINICAL TRIAL: NCT02894047
Title: Study of the Influence of the Expression of the Calcium-sensitive Receptor (CaSR) by Monocytes in the Synovial Liquid on Structural Alterations in Patients Diagnosed With Rheumatoid Arthritis in the Previous Two Years
Acronym: CASPER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2013_843_0014
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Arthritis, Rheumatoid
Keywords: calcium-sensitive receptor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood

INTERVENTIONS:
Biological: blood — measurement of CaSR expression levels on synovial fluid monocytes

SUMMARY:
Rheumatoid arthritis (RA) is the most frequent form of chronic inflammatory rheumatism in adults. The erosive damage influences the functional prognosis in patients with RA. At present, there are no sufficiently sensitive and specific predictive markers of erosive damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting in the Department of Rheumatology at Amiens University Hospital
* Age ≥ 18
* RA meeting the 2010 ACR/EULAR criteria
* Less than 2 years of RA progression
* Effusion in at least 1 joint

Exclusion Criteria:

* Inability to give informed consent
* Ongoing pregnancy
* Previous treatment with an anti-osteoporosis medication
* Intra-articular corticoid or hyaluronic acid injection in the previous 6 months
* Coagulation disorders preventing arthrocentesis
* Incarceration or legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients consulting in the Department of Rheumatology at Amiens University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
CaSR expression rate level on synovial monocytes | 1 year
  measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GOEB, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France